CLINICAL TRIAL: NCT02572765
Title: Evaluation of Splenic Metabolic Activity With 18FDG-PET in Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, prof. Giuseppe Lembo, Neuromed IRCCS
Other Study IDs: LMB05
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Total blood and serum

GROUPS / COHORTS (2):
- Normotensive: Normotensive subjects
  Interventions: Other: PET/CT scan
- Hypertensive: Hypertensive subjects
  Interventions: Other: PET/CT scan

INTERVENTIONS:
Other: PET/CT scan — PET/CT scan

SUMMARY:
The purpose of this study is to evaluate the splenic activation in hypertensive patients, as compared to normotensives, using FDG-PET/CT imaging. Moreover, the investigators will investigate whether the splenic metabolic activity relates to the expression of circulating inflammatory proteins (high-sensitivity C-reactive protein [hsCRP]), interleukin-1b (IL-1b), tumor necrosis factor-a (TNF-a) or to immune profiles of activated T cells.

ELIGIBILITY:
Inclusion Criteria:

* absence of prior cancer diagnosis or remission from cancer at the time of FDG-PET/CT imaging (from at least 6 months)
* age ≥ 30 and ≤ 85 years
* absence of acute cardio/cerebrovascular disease (myocardial infarction, stroke, transient ischemic attack, revascularization)
* absence of acute or chronic inflammatory or autoimmune disease
* diagnosis of presence/absence of hypertension, on the basis of documented medical history

Exclusion Criteria:

* diabetes
* atrial fibrillation
* use of anti-inflammatory drugs in the week preceding the FDG-PET/CT imaging
* chronic use of anti-inflammatory drugs

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients who will undergo FDG-PET/CT imaging of chest and abdomen in the Department of Nuclear Medicine of IRCCS Neuromed, accordingly to the following inclusion/exclusion criteria. All the enrolled patients must have an indication for FDG-PET/CT. Approximately 120 hypertensive and normotensive subjects of both genders (at least 45 per group, in order to have the appropriate statistical power) will be included in the study.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Splenic metabolic activity | At enrollment
  18FDG uptake in splenic tissue

SECONDARY OUTCOMES:
Circulating pro-inflammatory markers | At enrollment
  Serum levels of pro-inflammatory cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, (IS), Italy